CLINICAL TRIAL: NCT02471378
Title: In-Vitro Testing of Pregnancy Malaria Vaccine Candidates
Brief Title: Laboratory Evaluation of Pregnancy Malaria Vaccine Candidates/In-vitro Testing of Pregnancy Malaria Vaccine Candidates
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915147; 15-I-N147
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09-08

CONDITIONS: Malaria
Keywords: Assays; Women; Infected; Antibodies; Plasmodium Falciparum; Natural History
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women 15-25 years old: Malaria-infected pregnant Women

SUMMARY:
Background:

- Malaria is a disease that affects many people in African countries. It is caused by germs that are spread by mosquito bites. It can be fatal if not diagnosed and treated right away. Children younger than 5 and pregnant women are most at risk to get malaria. Researchers want to create a vaccine that will prevent malaria infection during pregnancy.

Objectives:

- To create a vaccine that will prevent malaria infection during pregnancy. To assess possible vaccines using in-vitro tests with parasites taken from pregnant women.

Eligibility:

- Pregnant women ages 15-25

Design:

* The study site is an area in Mali, West Africa.
* Participants:
* Will have blood drawn.
* Will give consent for the blood sample to be used for future research.
* May have a physical exam.
* Participants who have malaria or anemia will get treatment.

DETAILED DESCRIPTION:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences. Pregnancy malaria is associated with low birth weight (LBW), maternal anemia, and gestational hypertension; and both inflammation and the fetal response to infection may contribute to these poor outcomes. Pregnancy malaria (PM) is caused by P. falciparum-infected erythrocytes that bind to the placental receptor chondroitin sulfate A (CSA) and sequester in the placenta, where they cause disease and death for the mother and her offspring. Women become resistant to pregnancy malaria as they acquire antibodies that target surface proteins of placental parasites. Malaria vaccine candidates targeting the parasite s liver stage or blood stage may not protect pregnant women and their unborn children. The primary hypothesis in this study is that antibodies raised in animals against recombinant pregnancy malaria vaccine candidates will have a similar functional activity as naturally acquired antibodies. Up to 2492 malaria-infected pregnant women will be recruited into a cross sectional study that will be conducted in Ouelessebougou and neighboring districts, Mali. Women presenting for antenatal visit at the health centers in Ouelessebougou District will be enrolled. Samples collected from the women will be used in in-vitro assays to assess the functional activity of immunoglobulin G (IgG) raised against pregnancy malaria vaccine candidates as the primary outcome of this study. For our secondary outcomes, we will examine functional activity of naturally acquired antibodies specific to the vaccine candidates. Functional activity by IgG to vaccine candidates will be compared to the activity obtained with control proteins using appropriate statistical methods, including adjustment for possible confounders such as parasite density in the assay, to determine if the candidates elicit the type of immune response observed in naturally exposed population.

ELIGIBILITY:
* INCLUSION CRITERIA:

A study participant must satisfy the following criteria to be enrolled in this study:

* Pregnant women aged 15-25 years
* Able to provide consent for self
* Malaria positive by rapid diagnostic test (RDT)

EXCLUSION CRITERIA:

* Severe anemia defined as HGB<7 gr/dL, that may be worsened by 10 mL phlebotomy
* Conditions that in the judgment of the investigator could increase the risk to the volunteer
* Prior enrollment to the study during the same pregnancy

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women age 15-25 years presenting for antenatal consultations or delivery at health centers or hospital in Ouelessebougou and neighboring districts@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 7476 (Estimated)
Dates: Start 2015-07-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure of functional activity of animal IgG against vaccine candidates to block binding of fresh pregnancy malaria isolates to the placental receptor CSA | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fried, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ouelessebougou Clinical Research Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried M, Nosten F, Brockman A, Brabin BJ, Duffy PE. Maternal antibodies block malaria. Nature. 1998 Oct 29;395(6705):851-2. doi: 10.1038/27570. No abstract available. PMID 9804416
- [Background] Bordbar B, Tuikue-Ndam N, Bigey P, Doritchamou J, Scherman D, Deloron P. Identification of Id1-DBL2X of VAR2CSA as a key domain inducing highly inhibitory and cross-reactive antibodies. Vaccine. 2012 Feb 8;30(7):1343-8. doi: 10.1016/j.vaccine.2011.12.065. Epub 2012 Jan 5. PMID 22226864
- [Background] Fried M, Avril M, Chaturvedi R, Fernandez P, Lograsso J, Narum D, Nielsen MA, Oleinikov AV, Resende M, Salanti A, Saveria T, Williamson K, Dicko A, Scherf A, Smith JD, Theander TG, Duffy PE. Multilaboratory approach to preclinical evaluation of vaccine immunogens for placental malaria. Infect Immun. 2013 Feb;81(2):487-95. doi: 10.1128/IAI.01106-12. Epub 2012 Dec 3. PMID 23208604
- [Derived] Sharma A, Jenkins B, Akue A, Lambert LE, Orr-Gonzalez S, Thomas ML, Mahamar A, Diarra BS, Dicko A, Fried M, Duffy PE. Plasmodium falciparum in Aotus nancymaae: A New Model for Placental Malaria. J Infect Dis. 2022 Aug 26;226(3):521-527. doi: 10.1093/infdis/jiac096. PMID 35290467